CLINICAL TRIAL: NCT07382973
Title: Evaluation of Non-Thermal Plasma as an Innovative Strategy for Optimizing Post-Surgical Wound Treatment in Patients of Thyroid Surgery: An Ethical and Clinical Approach
Brief Title: Safety and Efficacy of NTP in Thyroid Surgery: Pilot Study on Morbidity Prevention and Adjuvant Oncological Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Nuclear Research - Mexico (Other)
Collaborators: Centro Medico Issemym (Other)
Responsible Party: Principal Investigator, Benjamín Gonzalo Rodríguez Méndez, Principal Investigator, National Institute of Nuclear Research - Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CISEI-201/25
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Diseases; Wound Healing; Thyroidectomy; Surgical Wound Infection
Keywords: Non-Thermal Plasma; Cold Plasma; Thyroid Surgery; Wound Healing; Postoperative Pain; Adjuvant Therapy; Surgical Bed Decontamination
MeSH Terms: conditions — Thyroid Diseases; Surgical Wound Infection; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Non-Thermal Plasma (NTP) (Experimental): The single experimental arm consists of patients undergoing total or partial thyroidectomy who receive a standardised treatment with Non-Thermal Plasma (NTP). This group is evaluated for surgical safety (nerve preservation/hemostasis) and oncological efficacy (residual disease control).
  Interventions: Device: Atmospheric Pressure Non-Thermal Plasma
- Standard Postoperative Care (Active Comparator): Participants randomized to this arm will receive the institution's current standard postoperative wound care following thyroid surgery. This includes routine surgical wound closure (sutures/staples) and standard dressing, without any application of non-thermal plasma. All other aspects of perioperative care, including pain management and follow-up visits, will follow standard institutional protocols.
  Interventions: Other: Standard Surgical Wound Care Protocol

INTERVENTIONS:
Device: Atmospheric Pressure Non-Thermal Plasma — Intraoperative and postoperative application of non-thermal plasma (NTP) generated via a 13.56 MHz Radiofrequency (RF) generator at 20 Watts. High-purity helium gas will be used as the precursor at a flow rate of 0.5 LPM. The plasma jet will be applied directly to the surgical bed (pre-closure) and the sutured incision (post-closure), maintaining a distance of 1-3 mm from the tissue. The dosage is standardized at 1 minute per linear centimeter of the incision.
  Arms: Treatment with Non-Thermal Plasma (NTP)
Other: Standard Surgical Wound Care Protocol — Standard surgical wound closure using conventional suturing techniques followed by the application of sterile dressings according to institutional protocols. No plasma treatment will be administered.
  Arms: Standard Postoperative Care

SUMMARY:
The goal of this clinical trial is to evaluate the therapeutic efficacy and safety of non-thermal plasma (NTP) as an adjuvant treatment for surgical bed decontamination and accelerated tissue repair in patients undergoing total thyroidectomy. The study aims to address the following objectives:

* Does the intraoperative application of NTP to the surgical bed and closed incision promote accelerated tissue regeneration compared to conventional postoperative care?
* Does NTP treatment reduce postoperative inflammatory response, pain intensity, and the incidence of site-specific complications (such as surgical site infection or seroma)?
* What is the safety profile of helium-based NTP in the cervical anatomical region regarding neighboring neurovascular structures?

Participants will be randomized into two arms:

1. The experimental group: Receiving a standardized application of helium-based NTP (at a frequency of 13.56 MHz) to the surgical bed prior to closure and subsequently to the sutured incision.
2. The control group: Receiving standard-of-care surgical wound management.

Clinical follow-up will include quantitative assessment of healing rates, pain scales (VAS), and biochemical or clinical markers of inflammation at scheduled intervals (Days 1, 7, 15, and up to 12 weeks post-surgery).

DETAILED DESCRIPTION:
This prospective study addresses the two most critical limitations of conventional thyroid surgery: collateral thermal damage to noble structures and the risk of microscopic residual disease in incidental carcinoma cases.

The investigation focuses on the application of non-thermal plasma (NTP), a state of matter that generates a controlled 'cocktail' of Reactive Oxygen and Nitrogen Species (RONS). Unlike conventional energy-based devices (laser or electrocautery), NTP operates at low temperatures, eliminating lateral thermal dispersion and carbonization, thus preserving the functional integrity of the recurrent laryngeal nerve and parathyroid glands.

The standardized NTP protocol is executed in two distinct phases:

1. Phase I (Hemostasis and Neuroprotection): Following thyroid gland resection, the surgical bed is exposed to a power density of 0.5 W/cm² for 8-10 minutes. This phase targets the carotid sheath and the tracheoesophageal groove to ensure immediate hemostasis and to modulate the inflammatory response through redox signaling, thereby preventing exuberant fibroplasia.
2. Phase II (Selective Oncological Ablation): In cases where incidental malignancy is suspected or confirmed, an additional re-exposure of 10-12 minutes is performed specifically on the resection micro-margins. This phase leverages the selective cytotoxicity of RONS, which induces mitochondrial dysfunction and apoptosis in neoplastic cells while sparing healthy surrounding tissue.

The study aims to correlate this two-phase intervention with three primary clinical pillars: a) Absolute surgical safety (0% complication rate in nerve paralysis and hypocalcemia). b) Oncological sterilization (undetectable Thyroglobulin levels <0.1 ng/dL at 6 months). c) High-fidelity tissue mimicry (evaluated via VSS and POSAS scales), hypothesizing that NTP-mediated redox modulation achieves superior cosmetic and functional outcomes compared to traditional photobiomodulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Diagnosis of thyroid pathology requiring total or subtotal thyroidectomy.
* Signed Informed Consent Form (ICF).
* Patients capable of complying with the 12-week follow-up schedule.

Exclusion Criteria:

* History of previous neck surgery or radiation therapy in the cervical area.
* Known history of keloid formation or hypertrophic scarring.
* Presence of active systemic or local infection at the time of surgery.
* Patients with implanted electronic devices (e.g., pacemakers or defibrillators) due to the use of RF-based plasma.
* Pregnancy or breastfeeding.
* Concurrent use of systemic corticosteroids or immunosuppressive drugs that may impair wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound re-epithelialization. | From day 0 (day of surgery) up to day 21.
  The number of days required for to achieve 100% skin closure of the surgical incision. Complete re-epithelialization is clinically defined as a fully closed wound without drainage, scabbing, or the need for dressings. Assessment will be performed by a blinded evaluator. Unit of measure: Days.

SECONDARY OUTCOMES:
Postoperative pain intensity. | At 2, 12, 24, 36, 48, and 72 hours, and on days 7 and 14 post-surgery.
  Patient-reported pain levels assessed using the Visual Analog Scale (VAS), where 0 represents "no pain" and 10 represents the worst imaginable pain. Unit of measure: VAS Score (0-10).
Incidence of surgical site complications. | From surgery through 28 days post-surgery.
  Total number of participants experiencing at least one postoperative complication, specifically: surgical site infection (SSI), wound dehiscence, hematoma, or seroma formation, as confirmed by clinical diagnosis. Unit of measure: Number of participants.
Long-term scar quality assessment. | At 12 weeks post-surgery.
  Objective evaluation of the scar using the Vancouver Scar Scale (VSS). The scale assesses four parameters: vascularity, pigmentation, pliability, and height. Total scores range from 0 to 13, with lower scores indicating better aesthetic and functional outcomes. Unit of measure: VSS Score (0-13).
Cumulative analgesic consumption. | First 48 hours post-surgery.
  Total amount of rescue analgesic medication (e.g., paracetamol or NSAIDs) required by the patient during the immediate postoperative period. This measure reflects the indirect impact of NTP on pain management. Unit of measure: Milligrams (mg) of medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Plasma Physics Laboratory, National Institute of Nuclear Research, Ocoyoacac, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Betancourt-Angeles M, Pena-Eguiluz R, Lopez-Callejas R, Dominguez-Cadena NA, Mercado-Cabrera A, Munoz-Infante J, Rodriguez-Mendez BG, Valencia-Alvarado R, Moreno-Tapia JA. Treatment in the healing of burns with a cold plasma source. Int J Burns Trauma. 2017 Dec 20;7(7):142-146. eCollection 2017. PMID 29348977
- [Background] Rodriguez-Mendez BG, Lopez-Callejas R, Mercado-Cabrera A, Pena-Eguiluz R, Valencia-Alvarado R, Betancourt-Angeles M, Berrones-Stringel G, Jaramillo-Martinez C. Harnessing Non-Thermal Plasma to Supercharge Recovery in Abdominal Surgeries: A Pilot Study. J Clin Med. 2024 Jan 11;13(2):408. doi: 10.3390/jcm13020408. PMID 38256546